CLINICAL TRIAL: NCT04692740
Title: A Pilot Study of Chlorambucil in Pre-treated Metastatic Pancreatic Adenocarcinoma Patients Bearing a Germ Line BRCA or Other DNA Defects Repair (DDR) Mutations.
Brief Title: Chlorambucil in Metastatic PDAC Patients Bearing a Germ Line DNA Defects Repair Mutations (SALE Trial)
Acronym: SALE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Michele Reni (Other)
Responsible Party: Sponsor-Investigator, Michele Reni, MD, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PACT29
Record Dates: First submitted 2020-12-30; First posted 2021-01-05 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: chlorambucil; BRCA mutations; DNA defect repair mutations
MeSH Terms: interventions — Chlorambucil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chlorambucil (Experimental)
  Interventions: Drug: Chlorambucil, Oral, 2 Mg

INTERVENTIONS:
Drug: Chlorambucil, Oral, 2 Mg — Eligible patients will be treated with Chlorambucil 6 mg/m2 daily p.o. for 42 consecutive days (weeks 1-6). After restaging, responder patients (complete or partial response) and those with stable disease will receive Chlorambucil 6 mg/m2 daily p.o for 14 consecutive days every 28 days until disease progression or unbearable toxicity, patient refusal or medical decision. Patients' clinical data will be collected pseudo-anonymously and a sequential identification code number will be assigned to each patient enrolled in the study.

SUMMARY:
The main objective of this trial is to explore the activity of chlorambucil, an alkylating agent commonly used in chronic lymphocytic leukemia treatment, in metastatic patients, gBRCA, including VUS, or DDR mutated, previously treated with a platinum-containing chemotherapy.

DETAILED DESCRIPTION:
Nowadays, treatment strategies for patients affected by metastatic pancreatic ductal adenocarcinoma (PDAC) are still very scant. Gemcitabine and fluoropyrimidine based chemotherapy regimens are standard I line chemotherapy. Recently, landmark genome-wide studies revealed the existence of a distinct subpopulation of PDAC with highly unstable genomic properties, due to mutations in DNA Damage Repair genes (DDR), in particular BRCA1/2 mutations. Germline mutations cause a deficiency in deoxyribonucleic acid (DNA) damage repair due to inhibition of DNA double-strand breaks repair by the mechanism of homologous recombination. Cancer cells rely on DNA repair to survive the damage induced by genotoxic stress and DNA repair enables cancer cells to accumulate genomic alterations that contribute to their aggressive phenotype. BRCA1/2 abrogation and homologous repair deficiency (HRD) confer sensitivity to DNA damage-inducing drugs, in particular those inflicting cytotoxic DNA crosslinks that interfere with DNA replication. The sensitivity of BRCA1/2-mutated tumors to platinum compounds has been validated in multiple pre-clinical and clinical studies. Nevertheless, similar lesions are induced by DNA-alkylating agents, which include mono-functional (e.g. mitomycin C) or bifunctional alkylators (e.g. chlorambucil). Small molecule inhibitors of poly(ADP-ribose) polymerase (PARP) have been recently developed and they showed an interesting activity and efficacy in breast, ovarian and pancreatic cancer tumors. Although platinum drugs and PARP inhibitors show initially good responses in the clinic, most patients acquire resistance to these drugs. Chlorambucil shows high selective toxicity against human cells and xenograft tumors with compromised BRCA1/2 function. Patients affected by metastatic ductal adenocarcinoma, pretreated with at least one previous platinum-based chemotherapy, will be treated with oral chlorambucil for 42 consecutive days After restaging, responder patients and those with stable disease will receive for 14 consecutive days every 28 days until disease progression (RECIST 1.1 criteria) or unbearable toxicity, patient refusal or medical decision.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed pancreatic adenocarcinoma
2. Age ≥ 18 years
3. ECOG PS 0-2
4. Stage IV disease
5. Identified genetic aberrations that are associated with homologous recombination deficiency (HRD)

   1. Cohort A: Documented mutation in gBRCA1 or gBRCA2 that is predicted to be deleterious or suspected deleterious
   2. Cohort B: BRCA1 or BRCA2 mutations that are considered to be of uncertain/unknown significance (VUS)
   3. Cohort C: Patients with other identified genetic aberrations that are associated with HRD
6. Adequate PFS during previous platinum-based chemotherapy for at least 4 months before progression
7. Screening laboratory values:

   Leukocytes > 3000/mmc Thrombocytes > 150000/mmc Hemoglobin > 10 g/dl Creatinine <2.0 times upper normal limit (unless normal creatinine clearance). Total bilirubin < 2.0 times upper normal limit (unless due to Gilbert's syndrome).

   Alanine aminotransferase (ALT) < 3.0 times upper normal limit.
8. Able to take oral medication
9. Progression during or after platinum-based chemotherapy
10. Other prior chemotherapy apart from first-line treatment for pancreatic cancer, are allowed, including maintenance treatment with PARP inhibitors
11. More than 2 weeks since prior chemotherapy end
12. Signed written informed consent
13. QTc <450 msec or QTc <480 msec for patients with bundle branch block

Exclusion Criteria:

1. Clinically significant cardiac disease including unstable angina, acute myocardial infarction within 6 months prior to screening, congestive heart failure, and arrhythmia requiring therapy, with the exception of extra systoles or minor conduction abnormalities
2. Active and uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy
3. Vaccination with vaccines called "live", since this treatment causes a drop of immunity defenses and a serious infection could result fatal.
4. History of seizure, head trauma and treatment with anti-epileptogenic drugs
5. Hypersensitivity to chlorambucil or to any excipients, in particular lactose
6. Recent radiotherapy (at least 4 weeks) or previous treatment with other cytotoxic agents
7. BRCA-mutated advanced pancreatic cancer who did not undergo maintenance with olaparib after platinum-based chemotherapy
8. Mismatch repair (MMR)/high levels of microsatellite instability (MSI-H), or high levels of tumor mutational burden (TMB) pancreatic cancer who did not undergo immunotherapy with pembrolizumab monotherapy or any other anti-PD1 agent
9. Concomitant PARP inhibitors therapy
10. Life expectancy less than 3 months, in the opinion of the investigator
11. Other past or current malignancy. Subjects who have been free of malignancy for at least 5 years, or have a history of completely resected non-melanoma skin cancer, or successfully treated in situ carcinoma are eligible
12. Symptomatic duodenal stenosis
13. CT contrast medium allergy and claustrophobia to RM investigation
14. Any significant medical condition laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study
15. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study
16. Any condition that confounds the ability to interpret data from the study
17. Any familiar, sociologic or geographic conditions that can potentially interfere with the adhesion to the protocol or to the follow-up
18. Pregnant or nursing. Adequate contraception is defined as oral hormonal birth control, intrauterine device, and male partner sterilization (if male partner is sole partner for that subject) and the double barrier method (condom or occlusive cap plus spermicidal agent).
19. Concurrent treatment with other experimental drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival evaluation | 6 months
  Evaluate the proportion of patients who are progression-free defined as progression according to RECIST 1.1 criteria or death. Progression free survival (PFS) is defined as the time between the date of registration and the date of documented radiological PD according to RECIST 1.1 criteria or death from any cause, whichever occurs first, or the date of last follow-up or last available tumour assessment if no further follow-up for disease progression is performed.

SECONDARY OUTCOMES:
Overall survival evaluation | 36 months
  Overall survival (OS) is defined as time between the date of registration and the date of death for any cause or the date they were last known to be alive
Radiological response rate | 6 months
  Radiological response evaluation by using RECIST 1.1 criteria
Biochemical response rate | 6 months
  Biochemical response evaluation by testing Ca19.9 marker
Drug safety | 6 months
  Drug toxicity evaluation by using appropriate SAE report form

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bailey P, Chang DK, Nones K, Johns AL, Patch AM, Gingras MC, Miller DK, Christ AN, Bruxner TJ, Quinn MC, Nourse C, Murtaugh LC, Harliwong I, Idrisoglu S, Manning S, Nourbakhsh E, Wani S, Fink L, Holmes O, Chin V, Anderson MJ, Kazakoff S, Leonard C, Newell F, Waddell N, Wood S, Xu Q, Wilson PJ, Cloonan N, Kassahn KS, Taylor D, Quek K, Robertson A, Pantano L, Mincarelli L, Sanchez LN, Evers L, Wu J, Pinese M, Cowley MJ, Jones MD, Colvin EK, Nagrial AM, Humphrey ES, Chantrill LA, Mawson A, Humphris J, Chou A, Pajic M, Scarlett CJ, Pinho AV, Giry-Laterriere M, Rooman I, Samra JS, Kench JG, Lovell JA, Merrett ND, Toon CW, Epari K, Nguyen NQ, Barbour A, Zeps N, Moran-Jones K, Jamieson NB, Graham JS, Duthie F, Oien K, Hair J, Grutzmann R, Maitra A, Iacobuzio-Donahue CA, Wolfgang CL, Morgan RA, Lawlor RT, Corbo V, Bassi C, Rusev B, Capelli P, Salvia R, Tortora G, Mukhopadhyay D, Petersen GM; Australian Pancreatic Cancer Genome Initiative; Munzy DM, Fisher WE, Karim SA, Eshleman JR, Hruban RH, Pilarsky C, Morton JP, Sansom OJ, Scarpa A, Musgrove EA, Bailey UM, Hofmann O, Sutherland RL, Wheeler DA, Gill AJ, Gibbs RA, Pearson JV, Waddell N, Biankin AV, Grimmond SM. Genomic analyses identify molecular subtypes of pancreatic cancer. Nature. 2016 Mar 3;531(7592):47-52. doi: 10.1038/nature16965. Epub 2016 Feb 24. PMID 26909576
- [Background] Pihlak R, Valle JW, McNamara MG. Germline mutations in pancreatic cancer and potential new therapeutic options. Oncotarget. 2017 Apr 20;8(42):73240-73257. doi: 10.18632/oncotarget.17291. eCollection 2017 Sep 22. PMID 29069866
- [Background] Rebelatto TF, Falavigna M, Pozzari M, Spada F, Cella CA, Laffi A, Pellicori S, Fazio N. Should platinum-based chemotherapy be preferred for germline BReast CAncer genes (BRCA) 1 and 2-mutated pancreatic ductal adenocarcinoma (PDAC) patients? A systematic review and meta-analysis. Cancer Treat Rev. 2019 Nov;80:101895. doi: 10.1016/j.ctrv.2019.101895. Epub 2019 Sep 6. PMID 31542591
- [Background] Golan T, Hammel P, Reni M, Van Cutsem E, Macarulla T, Hall MJ, Park JO, Hochhauser D, Arnold D, Oh DY, Reinacher-Schick A, Tortora G, Algul H, O'Reilly EM, McGuinness D, Cui KY, Schlienger K, Locker GY, Kindler HL. Maintenance Olaparib for Germline BRCA-Mutated Metastatic Pancreatic Cancer. N Engl J Med. 2019 Jul 25;381(4):317-327. doi: 10.1056/NEJMoa1903387. Epub 2019 Jun 2. PMID 31157963
- [Background] Tacconi EM, Badie S, De Gregoriis G, Reislander T, Lai X, Porru M, Folio C, Moore J, Kopp A, Baguna Torres J, Sneddon D, Green M, Dedic S, Lee JW, Batra AS, Rueda OM, Bruna A, Leonetti C, Caldas C, Cornelissen B, Brino L, Ryan A, Biroccio A, Tarsounas M. Chlorambucil targets BRCA1/2-deficient tumours and counteracts PARP inhibitor resistance. EMBO Mol Med. 2019 Jul;11(7):e9982. doi: 10.15252/emmm.201809982. Epub 2019 May 24. PMID 31273933